CLINICAL TRIAL: NCT00746018
Title: Evaluation of Thermal Spread Into the Interstitial Portion of the Fallopian Tubes Using the Ligasure Device at Time of Hysterectomy
Brief Title: Thermal Spread Into the Interstitial Portion of the Fallopian Tubes Using the Ligasure Device at Time of Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-092
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2017-07

CONDITIONS: Cervical Cancer; Ovarian Cancer; Uterine Cancer
Keywords: ovary; uterus; cervix; 08-092
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Uterine Neoplasms

ARMS (1):
- 1 (Experimental): The patients will already be undergoing a total hysterectomy with removal of the tubes and ovaries for a specific indication diagnosed or defined by their surgeon. If the patient is suitable to proceed by the surgeon, then he/she will perform a right salpingooophorectomy with the LigaSure devices.
  Interventions: Device: LigaSure vessel sealing system

INTERVENTIONS:
Device: LigaSure vessel sealing system — The investigators intend to enroll a total of 60 patients planned to undergo a total hysterectomy and bilateral salpingo-oophorectomy. There will be two techniques compared in this protocol. The first 30 patients will have the right tube removed with one application of the LigaSure. The LigaSure will be placed and the most proximal portion of the right fallopian tube adjacent to the uterine cornua and will be used to coagulate and cut the tube. The next 30 patients will have the tube ligated in the same fashion as group A however an additional step will be added once the fallopian tube has been removed. The LigaSure will be used to cauterize the remaining medial tissue on the cornua region of the uterus.

SUMMARY:
Some patients, specifically those with a diagnosed genetic mutation, will have their ovaries and fallopian tubes removed without removal of the uterus in an attempt to prevent ovarian and fallopian tube cancer from developing.

Anatomically the fallopian tubes are attached to the uterus and extend towards the ovaries. The fallopian tube tissue arises within the corner area of the uterus and occupies about 1cm of the uterine muscle wall.

The purpose of this study is to determine if the technique used to remove fallopian tubes only (without removal of the uterus) adequately removes or destroys all the fallopian tube cells that remain in the uterine muscle wall.

Currently, during the operation an instrument is used that burns the fallopian tube and allows it to be cut away from the uterus. The investigators do not know if this procedure successfully destroys all the fallopian tube cells within the uterus. Therefore, we will compare this single step procedure to a two step procedure. The two step procedure is to burn and cut the fallopian tube followed by an additional burning step, called cauterization at the top of the uterus. The investigators will assess if either or both of these procedures destroy the fallopian tube cells that may remain inside the uterine wall. This is important to determine since the goal is to remove the ovaries and all of the fallopian tubes in order to prevent future development of ovarian or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a non-emergent total hysterectomy with removal of the tubes and ovaries by the gynecologic service for benign or malignant conditions uterine, cervical or early ovarian cancer.
* Patients will undergo either a laparotomy, total laparoscopy or laparoscopically assisted vaginal hysterectomy
* Patients will be 21 years and older.

Exclusion Criteria:

* Patients with abnormal fallopian tubes seen preoperatively by radiologic exam or intraoperatively by visual inspection.
* Patients who are suspected to have fallopian tube cancer prior to their surgery
* Patients who have had prior pelvic radiation therapy
* Patients who are undergoing a Robotically Assisted procedure
* Patients who have had any type of prior tubal surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Abu-Rustum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Hysterectomy: The patients will already be undergoing a total hysterectomy with removal of the tubes and ovaries for a specific indication diagnosed or defined by their surgeon. If the patient is suitable to proceed by the surgeon, then he/she will perform a right salpingooophorectomy with the LigaSure devices.
Period: Overall Study
Arm/Group | Total Hysterectomy
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Hysterectomy
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 56 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: To Determine if the LigaSure Device, Which we Routinely Used for Removal of Tubes and Ovaries, is Effective at Destroying All Tubal Cells Comprising the Fallopian Tube Including Those Cells Within the Cornua of the Uterus.
Time Frame: conclusion of the study
Population: Data were not collected
Arm/Group | Total Hysterectomy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Total Hysterectomy
All-Cause Mortality (participants affected / at risk) | 4/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 34/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Hysterectomy (N=39)
Hyperglycemia (Metabolism and nutrition disorders) | 32
Hemoglobin (Blood and lymphatic system disorders) | 22
Hypoalbuminemia (Metabolism and nutrition disorders) | 18
Aspartate Aminotransferase (AST) Test (Investigations) | 7
Alanine Aminotransferase (ALT) Test (Investigations) | 6
Lymphopenia (Investigations) | 6
Hypokalemia (Metabolism and nutrition disorders) | 6
INR (Investigations) | 5
Platelets (Investigations) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 4
Alkaline phosphatase (Investigations) | 2
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2
Creatinine (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-04-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT00746018/Prot_SAP_000.pdf